CLINICAL TRIAL: NCT04884815
Title: An Operationally Seamless Phase 1/2/3 Study Consisting of a Safety and Dose-finding Phase 1/2 and Randomized, Open-label, Active-controlled Phase 3 to Evaluate UX701 AAV Gene Therapy in Adults With Wilson Disease
Brief Title: A Phase 1/2/3 Study of UX701 Gene Therapy in Adults With Wilson Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: UX701-CL301; 2020-005266-34 (EudraCT Number); 2022-502873-40-00 (Other: EU CT Number)
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Those responsible for reviewing MRI assessments, ophthalmology assessments, and analyzing liver biopsy samples will be double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Stage 1: UX701 Dose Level 1 (Experimental): Participants receive a single, peripheral intravenous (IV) infusion of UX701 at dose level 1.
  Interventions: Genetic: UX701
- Stage 1: UX701 Dose Level 2 (Experimental): Participants receive a single, peripheral IV infusion of UX701 at dose level 2.
  Interventions: Genetic: UX701
- Stage 1: UX701 Dose Level 3 (Experimental): Participants receive a single, peripheral IV infusion of UX701 at dose level 3.
  Interventions: Genetic: UX701
- Stage 1: UX701 Dose Level 4 (Experimental): Participants receive a single, peripheral IV infusion of UX701 at dose level 4.
  Interventions: Genetic: UX701
- Stage 2: UX701 at Selected Dose (Experimental): Participants randomized to UX701 receive a single, peripheral IV infusion of UX701 at the selected dose.
  Interventions: Genetic: UX701
- Stage 2: Standard of Care (SOC) to UX701 (Experimental): Participants randomized to SOC will continue their baseline SOC medications for 52 weeks, followed by a single, peripheral IV infusion of UX701 at the selected dose. Following UX701 administration, participants will be evaluated for modification of their SOC medications.
  Interventions: Genetic: UX701; Drug: Standard of Care (SOC)

INTERVENTIONS:
Genetic: UX701 — Nonreplicating, recombinant gene transfer vector
  Other Names: rivunatpagene miziparvovec
Drug: Standard of Care (SOC) — SOC treatment (i.e., copper chelators and/or zinc) administered according to standard regimens.
  Arms: Stage 2: Standard of Care (SOC) to UX701

SUMMARY:
The primary objectives of this study are to evaluate the safety of single IV doses of UX701 in patients with Wilson disease, to select the UX701 dose with the best benefit/risk profile based on the totality of safety and efficacy data and to evaluate the effect of UX701 on copper regulation.

DETAILED DESCRIPTION:
Stage 1 (Phase 1/2) is an open-label safety and dose-finding stage designed to evaluate the safety and efficacy of 4 dose levels of UX701 to establish initial safety of UX701 and select a safe and efficacious dose for further evaluation. Stage 2 (Phase 3) is a randomized, open-label, active-controlled stage to evaluate the safety and efficacy of UX701 using the dose selected in Stage 1. Stage 3 is a long-term follow-up stage designed to evaluate the safety, efficacy, and clinical benefit of UX701 for at least 5 years from the time of UX701 administration.

Participants who receive UX701 will receive premedication, prophylactic oral corticosteroids and immunomodulation therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of Wilson disease based on genetic confirmation of heterozygous or homozygous biallelic ATP7B mutation.
* Stable Wilson disease as evidenced by ongoing copper chelator (ie, penicillamine, trientine) and/or zinc therapy for at least 2 months at screening, with no medication or dose changes for at least 2 months at screening.
* Ongoing restriction of high copper containing foods for at least 2 months at Screening and continued through study participation.
* Willing and able to comply with all study procedures and requirements, including frequent blood collection, total urine collection over a 24-hour period, patient-reported outcome assessments, and long-term follow-up

Key Exclusion Criteria:

* Detectable pre-existing antibodies to the AAV9 capsid.
* Stage 1 only: History of copper chelator or zinc therapy noncompliance, in the Investigator's judgment, within 6 months prior to Screening.
* History of liver transplant.
* Active decompensated hepatic cirrhosis or history of hepatic encephalopathy.
* Significant hepatic inflammation as evidenced by laboratory abnormalities.
* Model for End-Stage Liver Disease (MELD) score > 13.
* Hemoglobin < 9 g/dL
* Presence of Stage 3 or higher chronic kidney disease based on estimated glomerular filtration rate < 60 mL/min/1.73 m2.
* Marked neurological deficit or compromise that, in the Investigator's opinion, would interfere with the subject's safety or ability to participate in the study.
* Moderate to severe depression, recent or active suicidal ideation with intent or suicidal behavior, psychosis, or unstable psychiatric illness.
* Known hypersensitivity to UX701 or its excipients, copper chelators, zinc, rituximab, tacrolimus, corticosteroids, or eculizumab that, in the Investigator's judgement, places the participant at increased risk for adverse events.
* Participation in another gene transfer study or use of another gene transfer product before or during study participation.
* Subjects with known hypersensitivity to amide-containing local anesthetics are excluded from participating in the optional liver biopsy substudy.

Note: Other protocol defined Inclusion/ Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2034-03 (Estimated)

PRIMARY OUTCOMES:
Stage 1: Incidence of Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs), Adverse Events of Special Interest (AESIs), Treatment-Related TEAEs, and Treatment-Related TESAEs | Up to Week 52
Stage 1: Change in 24-hour Urinary Copper Concentration from Baseline at Week 52 | Baseline, Week 52
Stage 1: Change in Total Copper from Baseline at Week 52 | Baseline, Week 52
Stage 1: Change in Ceruloplasmin-bound Copper from Baseline at Week 52 | Baseline, Week 52
Stage 1: Change in Ceruloplasmin from Baseline at Week 52 | Baseline, Week 52
Stage 1: Change in Non-Ceruloplasmin-bound Copper (NCC) from Baseline at Week 52 | Baseline, Week 52
Stage 1: Change in Free Copper from Baseline at Week 52 | Baseline, Week 52
Stage 1: Change in Ceruloplasmin Activity from Baseline at Week 52 | Baseline, Week 52
Stage 1: Percent Reduction in Standard of Care (SOC) Medication by Week 52 | Week 52
Stage 1: Number of Participants Who Discontinue SOC Medication by Week 52 | Week 52
Stage 1: Number of Consecutive Weeks off SOC Medication at Week 52 | Week 52
Stage 2: Change in 24-hour Urinary Copper Concentration from Baseline at Week 52, Evaluated for Superiority | Baseline, Week 52
Stage 2: Percent Reduction in SOC Medication by Week 52, Evaluated for Superiority | Week 52

SECONDARY OUTCOMES:
Stage 2: Change in Ceruloplasmin Activity Levels from Baseline at Week 52, Evaluated for Superiority | Baseline, Week 52
Stage 2: Number of Participants who Discontinue SOC Medication by Week 52 | Week 52
Stage 2: Change in FACIT-Fatigue Scale Score from Baseline at Week 52 | Baseline, Week 52
Stage 2: Change in Liver Copper Concentration Assessed by Liver Biopsy from Baseline at Week 52 | Baseline, Week 52

OTHER OUTCOMES:
Stage 2: Development of Anti-ATP7B Antibodies | Up to Week 104
Stage 2: Incidence of TEAEs, TESAEs, AESIs, Treatment-Related TEAEs, and Treatment-Related TESAEs | Up to Week 312

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (16):
- United States (11):
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Redwood City, California
  - University of California Davis, Sacramento, California
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia, Canada
- Portugal (2):
  - Centro Hospitalar Universitário Lisboa Norte, Lisbon, Lisbon District
  - Centro Hospitalar Universitário de São João, Porto, Porto District
- Hospital Universitario Vall d'Hebron - PPDS, Barcelona, Spain
- Kings College NHS Foundation, London, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to the rarity of Wilson Disease, individual patient data will not be shared in order to safeguard patient privacy. The study protocol and statistical analysis plan for this study will be available with the tabulated results once posted.

REFERENCES:
- See also: Ultragenyx Patient Advocacy/Wilson Disease Information — https://ultrarareadvocacy.com/wilson-disease-wd/
- See also: Ultragenyx Wilson Disease (WD) Research Study Opportunities — https://www.ultraclinicaltrials.com/WilsonDisease
- See also: Ultragenyx Transparency Commitment — https://www.ultragenyx.com/our-research/our-clinical-trial-transparency-commitment/